CLINICAL TRIAL: NCT00131781
Title: Cognitive Therapy Versus Supportive Therapy in Borderline Personality Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2000.230
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline personality disorder; Controlled trials; Cognitive Therapy; Supportive Therapy; suicide; impulsivity
MeSH Terms: conditions — Borderline Personality Disorder; Suicide; Impulsive Behavior | interventions — Cognitive Behavioral Therapy; Palliative Care

INTERVENTIONS:
Behavioral: Cognitive Therapy
Behavioral: Supportive Therapy

SUMMARY:
This is a randomised trial comparing cognitive therapy and supportive therapy administered along one year in borderline personality disorder. The follow-up is one year after treatments end.

The therapists were the same in the two groups. Patients received one session a week during six months and one session every two weeks during the next six months

DETAILED DESCRIPTION:
* Cognitive Therapy
* Structured session
* Conceptualization of the case with the patient
* Cognitive methods
* Guided discovery of the schemas
* Work on life-scenarios
* From scenarios to schemas
* Empathic confrontation to the schemas
* Building new schemas (Core belief work-sheet)
* Affective methods: role playing
* Interpersonal methods: counter transference issues
* Behavioral experiment
* Problem solving
* Consolidation methods
* Patients and therapists had manuals
* Supportive Therapy
* Therapist: active listening (face to face)
* Empathy
* Unconditional positive regard
* Reformulation and clarification
* Reflection of the patient's feelings
* Reassurance
* Therapist emphasizes the importance to ventilate problems
* Therapist answers some factual questions
* Therapist politely ignore or refuse requests for advice and directive attitudes
* Therapist demonstrates warmth and genuineness
* Patients and therapists had manuals

ELIGIBILITY:
Inclusion Criteria:

* DSM-4 DIBR >=8 (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Diagnostic inventory for borderline-revised)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2001-03

PRIMARY OUTCOMES:
Clinical Global Impression (CGI): Improvement (1-7): score 3 ( a little better) associated with a hopelessness scale score < 8 (this means that the suicide risk is low)

SECONDARY OUTCOMES:
CGI severity and improvement
Hamilton depression
Beck Depression Inventory
Hopelessness
Young: Schema Questionnaire II
Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition Personality Disorders Personality Questionnaire (SCID II PQ)
Minnesota Multiphasic Personality Inventory (MMPI) (minimult)
Eysenck: impulsivity scale
Checklist: impulsive risky behaviors
Quality of life
Handicap (Sheehan)
Time: Pre test, six months, post test and one year post treatment follow-up
Therapeutic relationship evaluation scale (patients and therapists)

CONTACTS AND LOCATIONS:
Overall Officials: Jean COTTRAUX, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital Pierre Wertheimer, Bron, France

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793